CLINICAL TRIAL: NCT05691205
Title: Identifying the Optimal Positive End-Expiratory Pressure Level to Ventilate Patients After Bilateral Lung Transplantation
Brief Title: Identifying Optimal PEEP After Lung Transplantation
Acronym: PEEP-LuTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Professor, Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0058711-U
Record Dates: First submitted 2023-01-11; First posted 2023-01-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant; Complications; Primary Graft Dysfunction
Keywords: Lung Transplantation; Primary Graft Dysfunction; Mechanical Ventilation; Positive End-Expiratory Pressure; Electrical Impedance Tomography
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEEP-LuTX (Experimental): Within 48h after LuTX we will evaluate the effects of three levels of PEEP (14>10>6 cmH2O) upon: - lung and chest wall mechanics, - intrapulmonary shunt fraction; - distribution of ventilation and perfusion; - gas exchange.
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — After a recruitment maneuver three levels of PEEP (14>10>6cmH2O) will be tested

SUMMARY:
Lung Transplantation (LuTX) is the curative treatment for selected patients with end-stage lung disease. Primary Graft Dysfunction (PGD), a specific form of respiratory failure occurring within the first 72 hours after graft reperfusion, represents the most common complication after LuTX.

Actual recommendation regarding management of mechanical ventilation of the lung graft immediately after LuTX are based only on opinion experts and not on clinical trials. Optimization of Positive End-Expiratory Pressure might contribute to both prevention and treatment of PGD.

In this interventional single-center non-pharmacological study (with medical device), in the immediate postoperative period of patients who are undergone LuTX, we will evaluate the effects of varying levels of PEEP upon: - lung and chest wall mechanics, - intrapulmonary shunt fraction; - distribution of ventilation and perfusion; - gas exchange.

The final aim is to find the optimal level of PEEP in this patient's cohort

ELIGIBILITY:
Inclusion Criteria:

* Recipient of LUTX
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Already undergone LUTX
* Major hemodynamic instability along the 24 hours following LUTX: systolic arterial pressure < 90 mmHg and/or heart rate > 120 beat/min and/or high dose vasopressor requirement (norepinephrine > 0.3 mcg/kg/min and/or epinephrine > 0.2 mcg/kg/min and/or dobutamine > 8mcg/kg/min)
* Documented post-LUTX endobronchial plasma leak requiring high levels of PEEP > 15 cmH2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Lung Compliance | Measurements at three PEEP levels during a decremental PEEP trial
  Identifying the level of PEEP associated to the best compliance

SECONDARY OUTCOMES:
Lung collapse&overdistension | Measurements at three PEEP levels during a decremental PEEP trial
  Identifying the level of PEEP associated to the lowest collapse&overdistension according to Electrical Impedance Tomography
Lung perfusion | Measurements at three PEEP levels during a decremental PEEP trial
  Identifying the level of PEEP associated to the most homogeneous distribution of lung perfusion according to Electrical Impedance Tomography
Intrapulmonary shunt | Measurements at three PEEP levels during a decremental PEEP trial
  Identifying the level of PEEP associated to the lowest intrapulmonary shunt level
Dead space | Measurements at three PEEP levels during a decremental PEEP trial
  Identifying the level of PEEP associated to the lowest dead space fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be shared with other researchers upon explicit request

REFERENCES:
- [Background] Diamond JM, Lee JC, Kawut SM, Shah RJ, Localio AR, Bellamy SL, Lederer DJ, Cantu E, Kohl BA, Lama VN, Bhorade SM, Crespo M, Demissie E, Sonett J, Wille K, Orens J, Shah AS, Weinacker A, Arcasoy S, Shah PD, Wilkes DS, Ware LB, Palmer SM, Christie JD; Lung Transplant Outcomes Group. Clinical risk factors for primary graft dysfunction after lung transplantation. Am J Respir Crit Care Med. 2013 Mar 1;187(5):527-34. doi: 10.1164/rccm.201210-1865OC. Epub 2013 Jan 10. PMID 23306540
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741